CLINICAL TRIAL: NCT06526377
Title: Phase II, Double Blind, Placebo Controlled, Randomized Study Examining Natrunix in Combination With Standard of Care in HLA-B27 Positive Subjects With Axial Spondyloarthritis
Brief Title: Natrunix in HLA-B27 Positive Subjects With Axial Spondyloarthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT064
Record Dates: First submitted 2024-06-15; First posted 2024-07-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Natrunix 400 mg Natrunix in Combination with Standard of Care (Experimental): This arm will have 40 subjects receiving Natrunix in Combination with Standard of Care in HLA-B27 Positive Patients with Axial Spondyloarthritis
  Interventions: Drug: Natrunix
- Placebo in combination with Standard of Care (Experimental): This arm will have 20 subjects receiving Placebo in Combination with Standard of Care in HLA-B27 Positive Patients with Axial Spondyloarthritis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natrunix — Natrunix is a monoclonal antibody preparation. Natrunix antibody is indistinguishable from a natural antibody isolated from a healthy human. Natrunix is expected to be the safest, most effective therapy for alleviating inflammatory pain and mitigating damage, mainly in the spine and sacroiliac joints, in AxSpA patients.
  Other Names: Vilamakitug
  Arms: Natrunix 400 mg Natrunix in Combination with Standard of Care
Drug: Placebo — Placebo
  Arms: Placebo in combination with Standard of Care

SUMMARY:
Double-blind, placebo-controlled, randomized trial of Natrunix in combination with Standard of Care in patients with Axial Spondyloarthritis

DETAILED DESCRIPTION:
This is Double-blind, placebo-controlled, randomized trial examining Natrunix in combination with Standard of Care. Qualified subjects will be consented and screened for study eligibility and enrollment. Enrolled subjects will be randomized in a 2:1 ratio to receive either 400 mg Natrunix or placebo. All subjects who enter the study must be on a stable background standard of care (SOC) that they were receiving for at least 8 weeks prior to study enrollment. Enrolled subjects must meet 2009 Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axial spondyloarthritis, be HLA-B27 positive, and have active disease as defined by a BASDAI score ≥4 or an ASDAS-CRP >2.1. Subjects will receive once weekly injection of Natrunix or placebo in addition to SOC for 12 weeks. The study will conclude after 12 weeks followed by a 12-week open label extension phase and one-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for HLA-B27 and have at least 2 additional SpA features OR Positive for HLA-B27 and has radiological evidence of sacroiliitis from either X-ray or MRI from patient's medical records.
2. Must have active disease at screening, according to either Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), with disease severity of ≥ 4 or ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score - C Reactive Protein) ≥ 2.1
3. Subject must be DMARD naive, including those who previously declined DMARD treatment options, OR previously discontinued DMARD treatment after initial trial of no more than 12 total weeks

Exclusion Criteria:

1. History of treatment with Natrunix
2. Have received any prior, or are currently receiving, treatment with opiates, csDMARDS, biologic DMARDs, JAK inhibitors, or other immunomodulatory agents for more than 12 weeks at any point prior to enrollment OR within 12 weeks prior to enrollment
3. Treatment with more than one csDMARD (such as methotrexate and sulfasalazine etc.) , biologic DMARD (such as Etanercept and Infliximab etc.), JAK inhibitor (such as Tofacitinib and Upadacitinib etc.), or any combination thereof prior to enrollment Currently requiring regular dosing regimen corticosteroids (excluding PRN dosing) Treatment with biologics that target CD20 (Rituximab or any other anti-CD20 antibody) prior to enrollment
4. Clinically significant laboratory abnormalities per PI's discretion
5. Positive for active HIV, hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Spondyloarthritis International Society (ASAS) criteria will be used to determine proportion of subjects achieving 40% Improvement (ASAS40 response) | At 12 weeks from Baseline
  In this study, sponsor will assess the safety and effectiveness of Natrunix (human antibody preparation) in combination with Standard of Care to determine the ASAS40 response rate. ASAS response is the measure of improvement in percentage of Axial Spondyloarthritis (AxSpA) disease. Patients who achieved at least 40% improvement on Assessment of Spondyloarthritis International Society (ASAS40) at week 12 will be considered as an ASAS40 responder for the primary analysis.

SECONDARY OUTCOMES:
Improvement/Deterioration in Patient's Global Assessment of Disease (PGA) Activity (using Numerical Rating Scale (NRS)) | At 12 weeks from Baseline
  A patient global assessment of Disease (PGA) will be administered to assess your overall treatment response and disease status in AxSpa. Subjects will be evaluated to estimate disease activity on a 0-10 scale where 10 is maximum worsening.
Pain assessment (using Numerical Rating Scale (NRS)) | At 12 weeks from Baseline
  Numerical Rating Scale for Pain (NRS) diary will be given to rate subject's pain from 0-10 (no pain to highest pain) for average pain and worst pain in past 24 hours.
Improvement/Deterioration in Function (Bath Ankylosing Spondylitis Functional Index (BASFI)) | At 12 weeks from Baseline
  The Bath Ankylosing Spondylitis Functional Index (BASFI) will be administered to assess the degree of subject's functional limitation. Questionnaires will ask the subjects the rate difficulty in daily activity on 0-10 scale where 0 is easy and 10 is impossible.
Improvement/Deterioration in inflammation (mean of questions 5 and 6 on the Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]) | At 12 weeks
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be administered to access subject's AxSpa. It to evaluate symptoms such as spinal pain, joint pain, morning stiffness duration/ severity, fatigue, and discomfort experienced. These symptoms will be assessed on scale of 0-10 where 0 is none and 10 is very severe.

OTHER OUTCOMES:
ASAS40 response | At Weeks 1, 3, 5, 8 and 10 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS40 indicates a ≥40% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS20 response | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation.
  ASAS20 indicates a ≥20% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS50 response | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS50 indicates a ≥50% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS70 response | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS70 indicates a ≥70% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
Improvement/deterioration in Patient's Global Assessment (PGA) of Disease Activity (using Numerical Rating scale (NRS)) both average and worst | At Weeks 1, 3, 5, 8 and 10 from Baseline
  A patient global assessment of Disease (PGA) will be administered to assess your overall treatment response and disease status in AxSpa. Subjects will be evaluated to estimate disease activity on a 0-10 scale where 10 is maximum worsening. Numerical Rating Scale for Pain (NRS) diary will be given to rate subject's pain from 0-10 (no pain to highest pain) for average pain and worst pain in past 24 hours.
Pain Assessment (using Numerical Rating Scale (NRS)) both average and worst | At Weeks 1, 3, 5, 8 and 10 from Baseline
  Numerical Rating Scale for Pain (NRS) diary will be given to rate subject's pain from 0-10 (no pain to highest pain) for average pain and worst pain in past 24 hours.
Improvement/deterioration in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be administered to access subject's AxSpa. It to evaluate symptoms such as spinal pain, joint pain, morning stiffness duration/ severity, fatigue, and discomfort experienced. These symptoms will be assessed on scale of 0-10 where 0 is none and 10 is very severe.
Improvement/deterioration in Bath Ankylosing Spondylitis Functional Index (BASFI) | At Weeks 1, 3, 5, 8 and 10 from Baseline
  The Bath Ankylosing Spondylitis Functional Index (BASFI) will be administered to assess the degree of subject's functional limitation. Questionnaires will ask the subjects the rate difficulty in daily activity on 0-10 scale where 0 is easy and 10 is impossible.
Improvement/deterioration in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  The enthesitis evaluation is performed based on 7 assessments:
  1. 1st costochondral joint left and right,
  2. 7th costochondral joint (left/right (LR)),
  3. posterior superior iliac spine LR,
  4. anterior superior iliac spine LR,
  5. iliac crest LR,
  6. 5th lumbar spinous process and
  7. proximal insertion of Achilles tendon left and right. Each anatomic site is graded for presence (1) or absence (0) of pain/tenderness. Total MASES score therefore ranges from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness).
Improvement/Deterioration in Tender Joint Count (TJC) | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  Tender Joint Count (TJC) will be used to assess the tenderness of your joints.
Improvement/Deterioration in Swollen Joint Count (SJC) | At Week 1, 3, 5, 8, 10, and 12 from Baseline
  Swollen Joint Count (SJC) will be used to assess the swelling of your joints.
Study Emergent Anterior Uveitis (AU) | At Weeks 0, 5 and 12 from Baseline
  The study emergent events of Anterior Uveitis will be documented and monitored in the study.
Improvement/Deterioration of Anterior Uveitis symptoms using Ocular Pain Assessment Survey (OPAS) | At 1, 3, 5, 8, 10, and 12 from Baseline
  The OPAS is a patient reported survey assessing eye pain location, eye pain intensity over the prior 24 hours and 2 weeks, eye pain impact on quality of life, eye pain aggravating/alleviating factors, eye pain associated factors, and associated non-eye pain intensity. Subjects will document the location of any eye pain on a diagram of the face and eyes, and the remaining questions will be answered utilizing either a 0-10 or 0%-100% scale as appropriate.
Improvement/Deterioration of Ankylosing Spondylitis Quality of Life (ASQoL) | At Weeks 1, 3, 5, 8, 10, and 12. from Baseline
  Ankylosing Spondylitis Quality of Life (ASQoL) is a valuable tool to access your quality of life living with ankylosing spondylitis. This includes answering 'Yes' or 'No' to the questions.
Evaluator's (Physician's) Global Assessment of Disease (EGA) | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  Evaluator's (Physician's) Global Assessment of Disease (EGA) will be administered to the subject by investigator to assess overall treatment response and disease status in AxSpA. It will be evaluated to estimate disease activity on a 0-10 scale where 10 is maximum worsening.
Improvement/Deterioration in response of Health Assessment Questionnaire Disability Index (HAQ-DI) | At Weeks 1, 3, 5, 8, 10, and 12 from Baseline
  Degree of disability was self-evaluated by participant using HAQ-DI.Assessment was made based on activities capable without any aids/devices. 20-question instrument assessed degree of difficulty person had in accomplishing tasks in 8 functional areas(dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0(indicated no difficulty)to 3(indicated inability to perform task in that area). Overall score computed as: sum of domain scores and divided by number of domains answered. Total possible score range:0-3 where 0=least difficulty and 3=extreme difficulty.
Improvement/Deterioration in inflammation (mean of questions 5 and 6 on the Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]) | At Weeks 1, 3, 5, 8 and 10 from Baseline
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be administered to access subject's AxSpa. It to evaluate symptoms such as spinal pain, joint pain, morning stiffness duration/ severity, fatigue, and discomfort experienced. These symptoms will be assessed on scale of 0-10 where 0 is none and 10 is very severe.
Number of subjects with increased dosage/new SOC medications | At Weeks 3, 8 and 12 from Baseline
  Number of subjects with increased dosage/new SOC medications will be compared between the treatment arms.
Number of subjects with reduced/discontinued SOC medications | At Weeks 3, 8 and 12 from Baseline
  Number of subjects with reduced/discontinued SOC medications will be compared between the treatment arms.
AEs and SAEs | 7 days from last dose
  All subjects who received study drug will be included in safety analysis. Safety analysis will be based on adverse events, vital signs, physical examinations, and clinical laboratory measurements. Adverse events will be grouped by System Organ Class (SOC) and Preferred Term (PT) within SOC according to the latest MedDRA coding dictionary.
Number of Participants with Clinically Significant Changes in Physical Examination Findings using the Physical Exam Assessment during the course of the study | up to 24 weeks
  Parameters assessed are below:
  General Appearance Head Eyes Ears Nose Mouth Throat Neck Lymph Nodes Pulmonary Cardiovascular Abdomen Skin Musculoskeletal Neurological
Number of Participants with Clinically Significant Changes in Vital Signs during the course of the study | up to 24 weeks
  Parameters assessed are below:
  Systolic Blood Pressure Diastolic Blood Pressure Pulse Body Temperature Peripheral Blood Oxygen Saturation Respiratory Rate
Number of participants with clinically significant abnormal value in laboratory test results which represent a change from pre-study values during the course of the study | up to 24 weeks
  Parameters assessed are below:
  Chemistry panel: Analysis to evaluate if you are in generally good health. Your body's electrolyte balance and the status/function of some of your internal organ systems will be assessed.
  Hematology Panel: Analysis to evaluate the levels of different types of blood cells present in your blood.
  Urinalysis: Subject's urine will be collected to analyze pH, protein, glucose, and blood cells (RBCs and WBCs).
ASAS40 response | At OLE weeks 17 and 24 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS40 indicates a ≥40% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS20 response | At OLE weeks 17 and 24 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS20 indicates a ≥20% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS50 response | At OLE weeks 17 and 24 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS50 indicates a ≥50% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
ASAS70 response | At OLE weeks 17 and 24 from Baseline
  ASAS response criteria consist of 4 domains that are of importance in assessing the improvement in signs and symptoms of patients with AS. These measures focus on AS disease activity, physical function, total spinal pain, and spinal stiffness/inflammation. ASAS70 indicates a ≥70% improvement in 3 of the 4 below domains and no worsening of 20% in the remaining domain.
  ASAS response criteria include improvements in each of the 4 domains: BASFI (Bath Ankylosing Spondylitis Functional Index) Patient Global Assessment of Disease Activity Total Spinal Pain Inflammation (Morning Stiffness)
Patient's Global Assessment of Disease Activity (using Numerical Rating Scale (NRS)) both average and worst | At OLE weeks 17 and 24 from Baseline
  A patient global assessment of Disease (using Numerical Rating Scale (NRS)) will be administered to assess your overall treatment response and disease status in AxSpa. Subjects will be evaluated to estimate disease activity on a 0-10 scale where 10 is maximum worsening.
Pain Assessment (using Numerical Rating Scale (NRS)) both average and worst | At OLE weeks 17 and 24 from Baseline
  Numerical Rating Scale for Pain (NRS) diary will be given to rate subject's pain from 0-10 (no pain to highest pain) for average pain and worst pain in past 24 hours.
Improvement/Deterioration in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | At OLE weeks 17 and 24 from Baseline
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be administered to access subject's AxSpa. It to evaluate symptoms such as spinal pain, joint pain, morning stiffness duration/ severity, fatigue, and discomfort experienced. These symptoms will be assessed on scale of 0-10 where 0 is none and 10 is very severe.
Improvement/Deterioration in Bath Ankylosing Spondylitis Functional Index (BASFI) | At OLE weeks 17 and 24 from Baseline
  The Bath Ankylosing Spondylitis Functional Index (BASFI) will be administered to assess the degree of subject's functional limitation. Questionnaires will ask the subjects the rate difficulty in daily activity on 0-10 scale where 0 is easy and 10 is impossible.
Improvement/Deterioration in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | At OLE weeks 17 and 24 from Baseline
  The enthesitis evaluation is performed based on 7 assessments:
  1. 1st costochondral joint left and right,
  2. 7th costochondral joint (left/right (LR)),
  3. posterior superior iliac spine LR,
  4. anterior superior iliac spine LR,
  5. iliac crest LR,
  6. 5th lumbar spinous process and
  7. proximal insertion of Achilles tendon left and right. Each anatomic site is graded for presence (1) or absence (0) of pain/tenderness. Total MASES score therefore ranges from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness).
Improvement/Deterioration in Tender Joint Count (TJC) | At OLE weeks 17 and 24 from Baseline
  Tender Joint Count (TJC) will be used to assess the tenderness of your joints.
Improvement/Deterioration in Swollen Joint Count (SJC) | At OLE weeks 17 and 24 from Baseline
  Swollen Joint Count (SJC) will be used to assess the swelling of your joints.
Study Emergent Anterior Uveitis (AU) | At OLE weeks 17 and 24 from Baseline
  The study emergent events of Anterior Uveitis will be documented and monitored in the study.
Improvement/Deterioration of Anterior Uveitis symptoms using Ocular Pain Assessment Survey (OPAS) | At OLE weeks 17 and 24 from Baseline
  The OPAS is a patient reported survey assessing eye pain location, eye pain intensity over the prior 24 hours and 2 weeks, eye pain impact on quality of life, eye pain aggravating/alleviating factors, eye pain associated factors, and associated non-eye pain intensity. Subjects will document the location of any eye pain on a diagram of the face and eyes, and the remaining questions will be answered utilizing either a 0-10 or 0%-100% scale as appropriate.
Improvement/Deterioration in Ankylosing Spondylitis Quality of Life (ASQoL) | At OLE weeks 17 and 24 from Baseline
  Ankylosing Spondylitis Quality of Life (ASQoL) is a valuable tool to access your quality of life living with ankylosing spondylitis. This includes answering 'Yes' or 'No' to the questions.
Evaluator's (Physician's) Global Assessment of Disease (EGA) | At OLE weeks 17 and 24 from Baseline
  Evaluator's (Physician's) Global Assessment of Disease (EGA) will be administered to the subject by investigator to assess overall treatment response and disease status in AxSpa. It will be evaluated to estimate disease activity on a 0-10 scale where 10 is maximum worsening.
Improvement/Deterioration in response of Health Assessment Questionnaire Disability Index (HAQ-DI) | At OLE weeks 17 and 24 from Baseline
  Degree of disability was self-evaluated by participant using HAQ-DI. Assessment was made based on activities capable without any aids/devices. 20-question instrument assessed degree of difficulty person had in accomplishing tasks in 8 functional areas(dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0(indicated no difficulty) to 3(indicated inability to perform task in that area). Overall score computed as: sum of domain scores and divided by number of domains answered. Total possible score range:0-3 where 0=least difficulty and 3=extreme difficulty.
Improvement/Deterioration in inflammation (mean of questions 5 and 6 on the Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]) | At OLE weeks 17 and 24 from Baseline
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be administered to access subject's AxSpa. It to evaluate symptoms such as spinal pain, joint pain, morning stiffness duration/ severity, fatigue, and discomfort experienced. These symptoms will be assessed on scale of 0-10 where 0 is none and 10 is very severe.
Number of subjects with increased dosage/new SOC medications | At OLE weeks 17 and 24 from Baseline
  Number of subjects with increased dosage/new SOC medications will be compared between treatment arms.
Number of subjects with reduced/discontinued SOC medications | At weeks 17 and 24 from Baseline
  Number of subjects with reduced/discontinued SOC medications will be compared between treatment arms.